CLINICAL TRIAL: NCT05567744
Title: Research Registry for Cerebral Autosomal Dominant Arteriopathy With Subcortical Infarcts and Leukoencephalopathy (CADASIL)
Brief Title: Registry for CADASIL
Status: Recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0827; A535100 (Other: UW Madison); SMPH/NEUROLOGY/NEUROLOGY (Other: UW Madison); Protocol Version 9/22/2022 (Other: UW Madison)
Record Dates: First submitted 2022-09-28; First posted 2022-10-05 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Cerebral Autosomal Dominant Ateriopathy With Subcortical Infarcts and Leukoencephalopathy
Keywords: CADASIL
MeSH Terms: conditions — CADASIL | interventions — Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CADASIL Registry Participants: Have a loved one or family member with CADASIL, or anyone with or at risk for CADASIL
  Interventions: Other: Registry

INTERVENTIONS:
Other: Registry — Registry

SUMMARY:
This study is being done in order to create a registry (list) of people interested in Cerebral Autosomal Dominant Arteriopathy with Subcortical Infarcts and Leukoencephalopathy (CADASIL) research. It may be that you have a family member or other loved one with CADASIL, or that you may have CADASIL or are at risk. Participation means that your name will be added to a list of people who will be invited to participate in future research studies on CADASIL. Participants must be 18 years or older, and will remain on the registry until they request to be removed.

DETAILED DESCRIPTION:
The purpose of this registry is to allow Dr. Jane Paulsen and her CADASIL research teams to contact individuals on the list who may fit a study's eligibility requirements. All individuals interested in CADASIL research who either have a family member or loved one, or are at risk themselves, are eligible to participate in this registry. Information collected as part of the registry will be used solely to determine potential participant's eligibility to participate research.

A patient registry is an organized system that uses observational study methods to collect uniform data (clinical and other) to evaluate specified outcomes for a population defined by a particular disease, condition, or exposure, and that serves a predetermined scientific, clinical, or policy purpose(s).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* have a loved one or a family member with CADASIL, or are at-risk for CADASIL themselves

Exclusion Criteria:

* Under 18 years of age

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study team will inform the lay community and professional society's memberships of the registry to assist with referrals for enrollment. Participants who are being contacted for other CADASIL research projects will be asked whether they would also like to enroll in the registry. Clinicians or other members of a patient's care team may also recruit participants out of their clinics.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2022-06-03 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
A Cerebral Autosomal Dominant Arteriopathy with Subcortical Infarcts and Leukoencephalopathy (CADASIL) Registry | Up to 20 years
  Create a list of persons willing to volunteer for CADASIL-related research to facilitate efficient recruitment.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Paulsen, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No